CLINICAL TRIAL: NCT07211997
Title: FebriDx® Pediatric Validation Study Protocol
Brief Title: FebriDx® Pediatric Validation Study
Status: Recruiting | Type: Observational
Sponsor: Lumos Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP-0021; 75A50124C000051 (Other Grant/Funding Number: BARDA)
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Acute Respiratory Infections (ARIs)
Keywords: Pediatric; Host immune response; Biomarkers; Point-of-Care; Myxovirus resistance protein A (MxA); C-reactive protein (CRP)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Respiratory and blood specimens will be retained for future testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Acute Respiratory Infection: Febrile pediatric patients (2-11 years) presenting to the emergency department, urgent care centers or primary care offices with suspected acute respiratory tract infection.
  Interventions: Device: FebriDx

INTERVENTIONS:
Device: FebriDx — Bacterial/Non-Bacterial Point-of-Care Assay that detects the presence of MxA and CRP in fingerstick blood

SUMMARY:
The primary objective of this study is to determine performance characteristics of the FebriDx® test in differentiating bacterial from non-bacterial etiology among febrile pediatric patients (2-11 years) presenting to the emergency department, urgent care center or primary care office with a suspected acute respiratory tract infection.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational, blinded study where children with suspected acute respiratory infection will undergo FebriDx® testing.

The primary outcome is the presence of a bacterial associated systemic host immune response related to a febrile acute respiratory tract infection, as compared to the reference standard of clinical adjudication as determined by a panel of pediatric experts using the Clinical Reference Algorithm that includes pathogen detection testing (e.g., bacterial culture, multiplex PCR) as well as measures of host immune response.

FebriDx is a rapid lateral flow immunoassay for the visual, qualitative, in vitro detection of elevated levels of host response proteins, Myxovirus resistance protein A (MxA) and C-reactive protein (CRP), directly from fingerstick blood.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by parent/guardian and Assent for ages 7-11 years
* Exhibit or report of a new onset measured temperature (oral or tympanic) of greater than or equal to 100.4°F/38°C within 3 days (72 hours) of enrollment
* Clinical suspicion for Acute Respiratory Infection beginning within 7 days before enrollment AND presents with at least one of the following new onset of symptoms: runny nose, nasal congestion, sore throat, cough, hoarse voice, shortness of breath / difficulty breathing

Exclusion Criteria:

* Unwilling to participate in 7-day follow-up or sign HIPAA waiver to obtain medical record if hospitalized
* Immunocompromised state or taking immunosuppressive or chemotherapeutic medications in the last 30 days (e.g. oral / inhaled steroids, Methotrexate, Cyclosporine, Chemotherapy, interferon therapy)
* Taking antibiotics or antiviral therapy in the last 14 days
* Received a live viral immunization in the last 14 days
* Clinical diagnosis of otitis media or recognizable viral syndrome (i.e., croup, varicella, stomatitis) at the time of enrollment
* Prior enrollment in the study

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients presenting to the emergency department, urgent care center or primary care office with a suspected acute respiratory tract infection
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Performance of the FebriDx® test | Day 1
  Positive Percent Agreement (PPA) and Negative Percent Agreement (NPA) of the FebriDx results in determining the presence of a bacterial associated systemic host immune response compared to the reference standard of clinical adjudication as determined by a panel of pediatric experts using the Clinical Reference Algorithm.
FebriDx Performance | Single visit
  Positive and negative percent agreement Presence of a bacterial associated systemic host immune response related to a febrile acute respiratory tract infection, as compared to the reference standard

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Avacare, Colton, California
  - PAS Research- Myrtle Avenue Pediatrics, Inc, Clearwater, Florida
  - PAS Research- Sandhill Pediatrics PA, Lutz, Florida
  - PAS Research, Tampa, Florida
  - Hometown Urgent Care, Huber Heights, Ohio
  - Hometown Urgent Care, Springfield, Ohio
  - PAS Research, Pittsburgh, Pennsylvania
  - Tribe, Charleston, South Carolina
  - Tribe- Parkside Pediatrics, Greenville, South Carolina
  - PAS Research, Edinburg, Texas